CLINICAL TRIAL: NCT04500340
Title: Test Anxiety: Pervasiveness, Link With Academic Achievement and Impact of Cognitive-behavioral Intervention in Its Reduction
Brief Title: Effectiveness of Cognitive Behavioral Therapy of Reduction of Test Anxiety
Acronym: GroupCBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Grants Commission (Other)
Responsible Party: Principal Investigator, Khem Raj Bhatta, Principal Investigator, University Grants Commission
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UGrantsCommission
Record Dates: First submitted 2020-07-18; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Test Anxiety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Cognitive Behavioral Therapy (Group CBT) (Experimental): Intervention Group will receive ten-session group CBT for test anxiety. Two sessions will be carried out each week.
  Interventions: Behavioral: Group CBT for test anxiety
- Control Group (No Intervention): The Control group will be waiting for the control group who will receive intervention if they demand after final assessment for outcome measure.

INTERVENTIONS:
Behavioral: Group CBT for test anxiety — The cognitive-behavioral therapy protocol developed by Flaxman, Bond & Keogh (2004) will be used as the intervention protocol. This protocol consists of 10 Sessions which are provided twice a week (each group will have 10 students).
  Arms: Group Cognitive Behavioral Therapy (Group CBT)

SUMMARY:
This study will evaluate the role of Group Cognitive Behavioral Therapy in test anxiety. The study participants will be psychology undergraduates with social work and psychology majors. The students will be selected among those who score three or more in Westside Test Anxiety Scale will participate in the study. Westside Test Anxiety will be used two weeks after completion of the group Cognitive Behavioral Therapy protocol (Flaxman, Bond & Keogh. 2004). The result will be analyzed using the t-test and Cohen's d.

ELIGIBILITY:
Inclusion Criteria:

* Those Studying Social work and Psychology as Major subjects, Those who have scored 3 and above in Westside Test Anxiety scale

Exclusion Criteria:

* Those scoring below 3 in Westside Test Anxiety Scale

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Westside Test Anxiety Scale (WTAS) | Change from Baseline Test Anxiety Scores after completion of Group Cognitive Behavioral Therapy ( after one and half month)
  The WTAS consists of 10 items, each using a Likert response scale where 1= "Never true" and 5= "always true. Total score is divided by 10 to obtain final scores. The total score ranges from one to five. Score of 1-2.9 is considered normal test anxiety and score of 3-5 is labelled as high test anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Khem R. Bhatta, Master, Principal Investigator — Tribhuvan University
Locations (1):
- Nepal Mega College and K and K International College, Kathmandu, Bagmati, Nepal